CLINICAL TRIAL: NCT04801680
Title: A Multicentric, Prospective Clinical Survey on Long Term Performance of an Acetabular Component in Primary Total Hip Arthroplasty
Brief Title: Mpact 3D Metal Cup PMS
Status: Recruiting | Type: Observational
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.023.01
Record Dates: First submitted 2020-12-16; First posted 2021-03-17 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Total Hip Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- Mpact 3d metal: Subjects, among those whose clinical condition makes them eligible for a primary total hip arthroplasty, will be invited to participate to the study during preoperative visit. The
  Interventions: Device: Mpact 3D metal cup

INTERVENTIONS:
Device: Mpact 3D metal cup — Subjects, among those whose clinical condition makes them eligible for a primary total hip arthroplasty, will be invited to participate to the study during preoperative visit. They'll receive the Mpact 3D metal cup device

SUMMARY:
Cementless fixation, with or without screw augmentation, has evolved during the past few decades as the preferred method for acetabular reconstruction. Although major improvements have been recorded with regard to clinical outcomes and survivorship, acetabular component loosening remains among the most common causes of failure and revision. Patient age, poor bone quality and conditions, such as osteonecrosis and dysplasia, have been observed to influence negatively long-term clinical results.

Initial stability is fundamental for survivorship of cementless cups. Prerequisites to achieve durable cementless cup fixation are close contact with viable native bone, primary mechanical stability and secondary bone integration. Press-fit techniques provide optimal conditions for bone ingrowth and fixation but research focused on cup material in order to improve primary stability. Pore size, bone-implant apposition, and material properties all influence bone ingrowth and long-term stability.

Biological ingrowth surfaces have become a standard prosthetic element in reconstructive hip surgery. A material's properties, three-dimensional architecture, and surface texture all play integral parts in its biological performance. Trabecular metal is an important new biomaterial that has been introduced to enhance the potential of biological ingrowth as well as provide a structural scaffold in cases of severe bone deficit. The continuity between the porous and solid parts has been specifically developed to overcome the limitations of the traditional porous coatings. In fact, the absence of an interface between the trabecular structure and the bulk material provides greater structural solidity and thus higher resistance to detachment and corrosion. Initial clinical applications have focused on bone restoration in tumor and salvage cases and in primary and revision reconstructive cases where the increased biological fixation would be of clinical benefit. However the bone ingrowth potential and mechanical integrity of this material offer exciting options for orthopedic reconstructive surgeons such as difficult THA cases, such as patients with high demands, subjects affected by severe hip conditions (i.e. osteonecrosis, dysplasia) or with extremely poor bone quality. Medacta Mpact 3D Metal cup, is an acetabular cup realized using the EBM (Electron Beam Melting) powder technology; this production method offers a high friction and scratch-fit feel for the initial stability, without the need of any additional coating. Moreover the 3D Metal structure creates a favorable environment for bone thus providing secondary fixation.

The aim of this study is to evaluate the long term clinical and radiological performance of MPact 3D Metal acetabular component.

ELIGIBILITY:
Inclusion Criteria:

* Those suffering from hip primary arthrosis, post-traumatic arthrosis, hip dysplasia or avascular necrosis of femoral head, rheumatic arthrosis
* Those aged between 18 and 75 years old at the surgery time
* those suitable to undergo to a primary total hip arthroplasty for whom the Mpact 3D Metal cup will be implanted (according to the label indication/contraindications)
* Patients who are willing and able to provide written informed consent for participation in the study. Written informed consent must be obtained prior to patient's surgery

Exclusion Criteria:

* Those with acute or chronic infection
* Those whose mental conditions may compromise their ability to provide informed consent to study participation, ability to complete questionnaires or complete 10-year follow-ups.
* Those suffered by severe deformation, at the discretion of surgeon
* Those suffered by osteoporosis
* Those with metabolic disorders that may involve bone metabolism for which cementless implants are contraindicated
* Those suffered by muscular atrophy or neuromuscular disease
* Those allergic to medical device material previewed for the surgery
* Those unable to give their consent to participate in the study or who do not want to participate
* Those whose functional recovery is compromised by

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: No sample size calculation has been performed; the number of patients has been defined according to the ODEP panel directive (Orthopaedic Data Evaluation Panel), for a long term post-marketing observational study. The number of patients is in line with long term observational study and considered sufficient to evaluate 10 years survival rate of the cup.
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2019-11-07 (Actual); Primary Completion 2032-12-07 (Estimated); Study Completion 2032-12-07 (Estimated)

PRIMARY OUTCOMES:
long term performance | 10 years
  Device survival will be assessed by Kaplan Meier curve

SECONDARY OUTCOMES:
Clinical performance | 3 months, 1, 5, 7 and 10 years after surgery
  Harris Hip Score collected during preoperative and follow-up visits. Harris Hip score scale correspond to 0-100 points. Results can be interpreted with the following: <70 = poor result; 70-80 = fair, 80-90 = good, and 90-100 = excellent.
Radiological performance | 3 months, 1, 5, 7 and 10 years after surgery
  standard x-ray exam performed preoperatively and postoperatively before discharge from hospital and during follow-up visits
Hip physical function after surgery | 3 months and 1, 5, 7 and 10 years after surgery
  HOOS-PS score collected during preoperative visit and follow-up visit. HOOS PS scale correspond to 100 (no difficulty) to 0 (extreme difficulty) scale.
Rate of complications | up to 10 years after surgery
  collection of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- IRRCCS Istituto Ortopedico Galeazzi, Milan, MI, Italy